CLINICAL TRIAL: NCT00485511
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Hydroxyurea in Spinal Muscular Atrophy
Brief Title: A Trial of Hydroxyurea in Spinal Muscular Atrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DOH96-TD-I-111-TM103
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea

SUMMARY:
Spinal muscular atrophy (SMA) is an autosomal recessive disorder in humans which results in the loss of motor neurons. It is caused by reduced levels of the survival motor neuron (SMN) protein as a result of loss or mutation of the SMN1 gene. SMN protein is encoded by two genes, SMN1 and SMN2, which essentially differ by an single nucleotide in exon 7. As a result, the majority of the transcript from SMN2 lacks exon 7. According to clinical severity, SMA was classified to three types, including type I, type II, and type III.

Drugs capable of modifying the transcription pattern of SMN2 to increase the full-length of SMN mRNA expression and the amount of SMN protein may have therapeutic effects for SMA patients. In order to test this hypothesis, we used EBV-transformed lymphoblastoid cell lines derived from the different types of SMA patients to screen the effect of various drugs on SMN2 gene expression. Hydroxyurea (HU) was found to be effective among the drugs we tested. HU is an effective therapeutic agent for patients with thalassemia and sickle cell disease which the toxicity is minimal and is well-tolerated and safely used in children. We had undergone a small-scaled 33 SMA patients randomized pilot trial (HU treatment for 8 weeks and then follow up drug-free 8 weeks) to evaluate the effect of HU in SMA patients and we got a promising preliminary data. We found that HU could significantly increase in the manual muscle testing scores at 4 weeks, and full-length SMN mRNA level in the 30mg/kg/day subgroup at 8 weeks relative to baseline, and it is safe under the dose 30mg/kg/day.

In this study, we plan to enroll 60 type II and III SMA patients and conduct a single-center, randomized, double-blind, placebo-controlled, prospective trial of two-year duration to evaluate the efficacy and safety of HU.The primary end points are the changes in full-length SMN expression, SMN protein, motor function and lung function in SMA patients. We also design a safety monitoring system to investigate the adverse effects and to assure the patients' safety. We hope we can find and prove the efficacy and safety of HU in SMA patients and set up a evaluating model for multi-center trials in the future.

ELIGIBILITY:
Inclusion Criteria:

* Sixty SMA patients fulfilled the diagnostic criteria of SMA as defined by the International SMA Consortium (Munsat, 1992), and all had homozygous deletion of SMN1 gene but carried SMN2 gene (Chang, 1995; 1997)
* The subjects shall each have the age older than 4 years.
* The subjects (if age > 20 years old) or their parents (if subject age < 20 years old) shall agree with the trial and have signed the informed consents.

Exclusion Criteria:

* The subjects shall not have hematological diseases, other severe systemic diseases and congenital anomalies except for SMA.
* The subjects shall not have severe perinatal asphyxia history.
* The subjects shall not be with respiratory assists.
* The subjects shall have normal hepatic and renal functions in the pre-trial examination.
* The subjects shall not have received operation with generalized anesthesia in past half a year.
* The subjects shall not have acceded to other clinical trials in past half a year.
* The subjects shall not get in this trial if they could not complete the course.

Min Age: 4 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuh Jyh Jong, MD, Principal Investigator — Vice President, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Grzeschik SM, Ganta M, Prior TW, Heavlin WD, Wang CH. Hydroxyurea enhances SMN2 gene expression in spinal muscular atrophy cells. Ann Neurol. 2005 Aug;58(2):194-202. doi: 10.1002/ana.20548. PMID 16049920